CLINICAL TRIAL: NCT01108172
Title: A Virtual Ward to Reduce Readmissions After Hospital Discharge
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Toronto Central Local Health Integration Network (Unknown); Ontario Ministry of Health and Long Term Care (Other Government); Toronto Central Community Care Access Centre (Other); Women's College Hospital (Other); University Health Network, Toronto (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Irfan Dhalla, Staff Physician & Scientist, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 216852-PHE-CEAJ-25173
Record Dates: First submitted 2010-04-13; First posted 2010-04-21 (Estimated); Last update posted 2013-12-09 (Estimated); Status verified 2013-12

CONDITIONS: Acute Disease
MeSH Terms: conditions — Acute Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Active Comparator)
  Interventions: Other: Usual care
- Virtual Ward (Experimental)
  Interventions: Other: Virtual Ward

INTERVENTIONS:
Other: Virtual Ward — A multidisciplinary team to optimize medical and social care for patients residing in their own homes
  Arms: Virtual Ward
Other: Usual care — The usual care provided to patients after discharge from hospital
  Arms: Usual Care

SUMMARY:
The purpose of this study is to see whether a Virtual Ward reduces readmissions after hospital discharge.

DETAILED DESCRIPTION:
We will conduct a pragmatic, randomized controlled trial to evaluate a new model of care for high-risk medical patients after discharge from hospital. This new model of care has two key elements. First, we will use the LACE index (see citation below for details) to identify patients who are at high risk of readmission or death after hospital discharge. These patients will be randomized to either the Virtual Ward or usual care on the day of discharge. Although patients being cared for in the Virtual Ward will reside at home, they will benefit from a hospital-like interdisciplinary team, a shared set of notes, a single point of contact, round-the-clock physician availability and increased co-ordination of specialist, primary and home-based community care for several weeks after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Discharge from medical service
* LACE score greater than or equal to 10
* Age greater than or equal or 18
* Resident in Toronto Central Local Health Integration Network catchment area
* Patient or designate able to speak English well enough for follow up telephone calls

Exclusion Criteria:

* Previously enrolled in study
* Discharged to a rehabilitation or complex continuing care facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1928 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Composite of readmission to hospital or death. | 30 days after hospital discharge
  A binary outcome variable for each patient, representing either readmission to hospital or death within 30 days of hospital discharge. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.

SECONDARY OUTCOMES:
Composite of readmission or death | 90 days after discharge
  A binary outcome variable for each patient, representing either readmission to hospital or death within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Composite of readmission or death | 6 months after discharge
  A binary outcome variable for each patient, representing readmission to hospital within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Composite of readmission or death | One year after discharge
  A binary outcome variable for each patient, representing either readmission to hospital or death within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Emergency department visits | 30 days after discharge
  A binary outcome variable for each patient, representing an emergency department visit within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Emergency department visits | 90 days after discharge
  A binary outcome variable for each patient, representing an emergency department visit within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Emergency department visits | 6 months after discharge
  A binary outcome variable for each patient, representing an emergency department visit within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Emergency department visits | One year after discharge
  A binary outcome variable for each patient, representing an emergency department visit within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Long-term care admission | 30 days after discharge
  A binary outcome variable for each patient, representing a long-term care admission within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Long-term care admission | 90 days after discharge
  A binary outcome variable for each patient, representing a long-term care admission within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Long-term care admission | 6 months after discahrge
  A binary outcome variable for each patient, representing a long-term care admission within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Long-term care admission | One year after discharge
  A binary outcome variable for each patient, representing a long-term care admission within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Death | 90 days after discharge
  A binary outcome variable for each patient, representing death within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences
Death | 6 months after discharge
  A binary outcome variable for each patient, representing death within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences
Death | One year after discharge
  A binary outcome variable for each patient, representing death within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences
Death | 30 days after discharge
  A binary outcome variable for each patient, representing death within the time periods noted above. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences
Composite of readmission to hospital or death. | One year after discharge
  Time to the composite outcome of either readmission to hospital or death. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Data will be censored on the date of the last follow up (i.e., 30 days, 90 days or 6 months). Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Readmission | One year after discharge
  Time to readmission to hospital. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Data will be censored on the date of the last follow up (i.e., 30 days, 90 days or 6 months), or on death. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Emergency department visits | One year after discharge
  Time to emergency department visit. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Data will be censored on the date of the last follow up (i.e., 30 days, 90 days or 6 months), or on readmission or death. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Long-term care admission | One year after discharge
  Time to long-term care admission. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Data will be censored on the date of the last follow up (i.e., 30 days, 90 days or 6 months), or on death. Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.
Death | One year after discharge
  Time to death. A research assistant blinded to the assignment will ascertain this information via telephone using a standardized script. Data will be censored on the date of the last follow up (i.e., 30 days, 90 days or 6 months). Second, we may also ascertain this information by linking the data we collect to administrative databases housed at the Institute for Clinical Evaluative Sciences.

CONTACTS AND LOCATIONS:
Overall Officials: Irfan Dhalla, MD, MSc, Principal Investigator — St. Michael's Hospital/University of Toronto
Locations (5):
- Canada (5):
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Central Community Care Access Centre, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario

REFERENCES:
- [Background] van Walraven C, Dhalla IA, Bell C, Etchells E, Stiell IG, Zarnke K, Austin PC, Forster AJ. Derivation and validation of an index to predict early death or unplanned readmission after discharge from hospital to the community. CMAJ. 2010 Apr 6;182(6):551-7. doi: 10.1503/cmaj.091117. Epub 2010 Mar 1. PMID 20194559
- [Derived] Dhalla IA, O'Brien T, Morra D, Thorpe KE, Wong BM, Mehta R, Frost DW, Abrams H, Ko F, Van Rooyen P, Bell CM, Gruneir A, Lewis GH, Daub S, Anderson GM, Hawker GA, Rochon PA, Laupacis A. Effect of a postdischarge virtual ward on readmission or death for high-risk patients: a randomized clinical trial. JAMA. 2014 Oct 1;312(13):1305-12. doi: 10.1001/jama.2014.11492. PMID 25268437